CLINICAL TRIAL: NCT05167604
Title: Utility of ctDNA In Predicting Whether Giving Adjuvant Chemotherapy In Patients With Stage IB-IIA Resected Non-small Cell Lung Cancer: A Prospective Cohort Study
Brief Title: Clinical Value of MRD Monitoring for Adjuvant Therapy in Postoperative NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 777436
Record Dates: First submitted 2021-11-05; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Next-Generation Sequencing; Chemotherapy, Adjuvant; Neoplasm, Residual; Circulating Tumor DNA
Keywords: non-small cell lung cancer; next-generation sequencing; adjuvant chemotherapy; minimal residual disease; circulating tumor DNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual | interventions — Adjuvants, Pharmaceutic; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Circular DNA from the blood samples of NSCLC patients before and after adjuvant chemotherapy were collected and examined by NGS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MRD-positive Cohort: ctDNA positivity in pretreatment and posttreatment plasma samples was defined by accessing the presence of one or more mutations identified in match tumor samples. A mutation was considered present when at least one consensus read contained the mutation and passed the local polishing pipeline. The MRD positive cohort was randomly divided into two groups, one group for interventional treatment and the other group for observation.
  Interventions: Drug: Adjuvants, Pharmaceutic
- MRD-negative Cohort: ctDNA negative in pretreatment and posttreatment plasma samples was defined by accessing the presence of no mutation identified in match tumor samples. According to the clinical prognostic characteristics of the MRD negative group, the clinician decides to observe or treat.
  Interventions: Drug: Adjuvants, Pharmaceutic

INTERVENTIONS:
Drug: Adjuvants, Pharmaceutic — Patients with stage IB-IIA NSCLC after curative surgery were treated with adjuvant chemotherapy. The blood samples of the patients before and after adjuvant chemotherapy will be collected to examine the MRD status
  Other Names: adjuvant chemotherapy

SUMMARY:
This clinical trial aims to explore the minimal residual disease (MRD) status of early NSCLC after curative surgery and the clinical outcomes of adjuvant chemotherapy. Next-generation sequencing technique will be used to examine the circulating tumor DNA (ctDNA) from MRD of 150 postoperative patients with stage IB-IIA NSCLC who received adjuvant chemotherapy.

DETAILED DESCRIPTION:
Minimal residual disease (MRD) refers to the small number of malignant cells that remain after curative treatments (curative intent surgical resection, radiotherapy, and/or chemotherapy). MRD is common in patients with blood cancer, and is known to be associated with recurrence and poor prognosis. Recent studies also reported that MRD-negative in postoperative solid tumors such as colorectal/colon cancer and breast cancer is associated with better survival outcomes. However, the clinical values of MRD monitoring for adjuvant therapy in postoperative NSCLC remain inadequate.

Circulating tumor DNA (ctDNA), a type of cell-free DNA, refers to the DNA fragments that are derived from tumor cells and circulate in the blood. Recently, next-generation sequencing (NGS) was successfully applied to monitor NPM1, RUNX1 and FLT3 mutations in multiple myeloma. Thus, NGS technique is a promising tool for sensitive MRD monitoring, which provides the ctDNA profiling from MRD, and then provides future decision-making treatment for postoperative NSCLC patients. Thus, this clinical study aims to monitor the ctDNA status of MRD, and to explore the clinical value of MRD monitoring in decision-making adjuvant therapy for patients with stage IB-IIA NSCLC after curative surgery.

A total of 150 patients with primary curable stage IB-IIA NSCLC will be recruited in this clinical trial. The following samples will be collected from each patient including 1) preoperative blood samples; 2) surgical tissue samples; 3) blood samples 3-7 days after surgery; 4) blood samples every 3-6 month during adjuvant chemotherapy; and 5) white blood control samples. In addition, demographic and tumor characteristics of the patients will be collected for subsequent analysis, including age, sex, tumor stage, pathological stage, disease couse time, PS score, etc. NGS will be used to analyze the whole exons of potential driver genes to obtain the MRD status. Statistical analyses will be performed to analyze the survival outcomes of MRD-positive and MRD-negative group and to explore the clinical value of MRD monitoring for adjuvant therapy in postoperative NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Histological diagnosis of primary NSCLC
* Patients received curative surgery for primary NSCLC
* Tumor stage IB-IIA after curative-intent surgical resection
* ECOG score: 0-1
* Participant is willing to use an acceptable form of contraception during the study.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* The patient has received neoadjuvant therapy, including radiotherapy and chemotherapy, targeted therapy and immunotherapy
* Patients are unwilling or unable to receive the curative-intent resection
* Patients have or have had history of malignant tumor
* Patients who suffer from severe uncontrolled disease that require systemic treatment or considered unsuitable for participating this trial due to other reasons by the investigator
* Patients with severe gastrointestinal dysfunction, cardiac dysfunction, interstitial lung disease, etc.
* Laboratory test results showed inadequate bone marrow or organ function
* Blood transfusion during or within 2 weeks before the surgery
* History of alcohol abuse or drug overdose
* Pregnant or breastfeeding women
* Patients who are currently or have participated in any other anti-tumor clinical trials
* Inadequate baseline data, such as preoperative and postoperative blood samples (Lack of 2 consecutive blood test or a total of 3 blood samples), surgical tumor tissues, and ctDNA test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patents with histologically confirmed primary NSCLC, stage IB-IIA, aged 18-70 years
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | 3 years
  DFS defined as the time from randomization to occurrence of any of the following events, whichever occurs first:
  Locoregional recurrence or distant metastases as determined by an independent central radiology assessment.
  Occurrence of the second primary (same or other) cancer as determined by an independent central radiology assessment.
  Death from any cause. Loss to follow-up is censored.

SECONDARY OUTCOMES:
ctDNA status | Through study completion, up to 5 years
  Change of Circulating tumor DNA (ctDNA) status (every 3 months)
TEAE | Through study completion, up to 3 years
  Occurrence of treatment emergent adverse event (TEAE)
IMP | Through study completion, up to 3 years
  Occurrence of dose reduction and discontinuation of IMP due to a TEAE
Overall survival | 3 years and 5 years
  Follow-up of the patients will be conducted to analyze 3-year and 5-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Principal Investigator — Department of Thoracic Surgery, Tangdu Hospital, the Fourth Military Medical University
Locations (1):
- The Second Affiliated The Second Affiliated Hospital of Air Force Medical University (Tangdu Hospital), Xi'an, Baqiao, China

IPD SHARING:
Plan to Share IPD: No
The trial is recruiting patients

REFERENCES:
- [Result] Rolfo C, Castiglia M, Hong D, Alessandro R, Mertens I, Baggerman G, Zwaenepoel K, Gil-Bazo I, Passiglia F, Carreca AP, Taverna S, Vento R, Santini D, Peeters M, Russo A, Pauwels P. Liquid biopsies in lung cancer: the new ambrosia of researchers. Biochim Biophys Acta. 2014 Dec;1846(2):539-46. doi: 10.1016/j.bbcan.2014.10.001. Epub 2014 Oct 16. PMID 25444714
- [Result] Chin RI, Chen K, Usmani A, Chua C, Harris PK, Binkley MS, Azad TD, Dudley JC, Chaudhuri AA. Detection of Solid Tumor Molecular Residual Disease (MRD) Using Circulating Tumor DNA (ctDNA). Mol Diagn Ther. 2019 Jun;23(3):311-331. doi: 10.1007/s40291-019-00390-5. PMID 30941670
- [Result] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Result] Tie J, Cohen JD, Wang Y, Christie M, Simons K, Lee M, Wong R, Kosmider S, Ananda S, McKendrick J, Lee B, Cho JH, Faragher I, Jones IT, Ptak J, Schaeffer MJ, Silliman N, Dobbyn L, Li L, Tomasetti C, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating Tumor DNA Analyses as Markers of Recurrence Risk and Benefit of Adjuvant Therapy for Stage III Colon Cancer. JAMA Oncol. 2019 Dec 1;5(12):1710-1717. doi: 10.1001/jamaoncol.2019.3616. PMID 31621801
- [Result] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Result] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Result] Olsson E, Winter C, George A, Chen Y, Howlin J, Tang MH, Dahlgren M, Schulz R, Grabau D, van Westen D, Ferno M, Ingvar C, Rose C, Bendahl PO, Ryden L, Borg A, Gruvberger-Saal SK, Jernstrom H, Saal LH. Serial monitoring of circulating tumor DNA in patients with primary breast cancer for detection of occult metastatic disease. EMBO Mol Med. 2015 Aug;7(8):1034-47. doi: 10.15252/emmm.201404913. PMID 25987569
- [Result] Sausen M, Phallen J, Adleff V, Jones S, Leary RJ, Barrett MT, Anagnostou V, Parpart-Li S, Murphy D, Kay Li Q, Hruban CA, Scharpf R, White JR, O'Dwyer PJ, Allen PJ, Eshleman JR, Thompson CB, Klimstra DS, Linehan DC, Maitra A, Hruban RH, Diaz LA Jr, Von Hoff DD, Johansen JS, Drebin JA, Velculescu VE. Clinical implications of genomic alterations in the tumour and circulation of pancreatic cancer patients. Nat Commun. 2015 Jul 7;6:7686. doi: 10.1038/ncomms8686. PMID 26154128